CLINICAL TRIAL: NCT06624839
Title: A PRe-pOsT Interventional Study Evaluating Gardasil Nine-valent Human Papilloma Virus (HPV) Vaccine Humoral and Cellular Immune Responses in People With or Without HIV
Brief Title: Evaluating Gardasil HPV Vaccine Humoral and Cellular Immune Responses in People With and Without HIV
Acronym: PROTECT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00109701
Record Dates: First submitted 2024-07-30; First posted 2024-10-03 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Human Papilloma Virus; Anal Dysplasia; HIV
MeSH Terms: interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- People born male with current or past exposure to androgen blockers or estrogen (BM-EABE) (Experimental): One dose of human papillomavirus (HPV) vaccine, 9-valent (Gardasil9) will be administered on Day 0, Month 2, and Month 6
  Interventions: Biological: Human papillomavirus (HPV) vaccine, 9-valent
- HIV Negative BM-EABE or HIV Negative men who had sex with a person with a penis (MSPP) (Active Comparator): One dose of human papillomavirus (HPV) vaccine, 9-valent (Gardasil9) will be administered on Day 0, Month 2, and Month 6
  Interventions: Biological: Human papillomavirus (HPV) vaccine, 9-valent

INTERVENTIONS:
Biological: Human papillomavirus (HPV) vaccine, 9-valent — 0.5 ml intramuscular injection
  Other Names: Gardasil9

SUMMARY:
This is a phase 2, open-label study to assess the immunogenicity of the 9-valent human papillomavirus (HPV) recombinant vaccine (Gardasil9) in people born male with current or past exposure to androgen blockers or estrogen (BM-EABE). Investigators will enroll BM-EABE with HIV and HIV negative controls (BM-EABE or men who have sex with a person with a penis (MSPP)) and administer Gardasil9 at timepoints Day 0, Month 2, and Month 6. The immune response to the vaccine will be analyzed at Month 7 (1 month following the final vaccine dose).

DETAILED DESCRIPTION:
This will be a phase 2, open-label study to assess the humoral and cellular immune response to the FDA-approved 9-valent HPV recombinant vaccine in people born male with current or past exposure to androgen blockers or estrogen (BM-EABE). At baseline, BM-EABE with HIV, HIV negative controls (BM-EABE or men who have sex with a person with a penis (MSPP)) will provide blood samples and anal swabs for evaluation of HPV immunity, anal HPV and anal dysplasia. All participants will undergo a 3-dose vaccine series of the Gardasil vaccine (at Day 0, Month 2 and Month 6). Participants will then return one month after completion of third vaccine (Month 7) to provide repeat blood samples and anal swabs. Samples will be compared pre and post vaccination and in-between participants based on HIV and exposure to androgen blockers or estrogen (EABE).

Any participant with human papillomavirus 16 (HPV16) and/or anal dysplasia on anal cytology at any point will be referred to high-resolution anoscopy (HRA) for clinical management. Anal biopsies will be procured from different pathology laboratories - after clinical evaluation has been complete - for research analysis, including confocal microscopy. Those who had anal dysplasia at study entry will undergo repeat HRA, as clinically indicated, and will have an optional study visit following their repeat HRA to provide blood draw and anal swabs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older and 70 years old or younger
* Able to provide informed consent
* Denies history of prior HPV vaccination with Gardasil9 (receipt of HPV vaccination other than Gardasil9 such as the bivalent or the quadrivalent HPV vaccine will be allowed) or unsure of vaccination status and born before 2003
* Born Male

For Test group: HIV-positive people born male with current or past exposure to androgen blockers or estrogen (BM-EABE)

* Living with HIV
* Current or past exposure to androgen blockers or estradiol

For Control group: HIV-negative Control

* HIV negative
* Either: Current or past exposure to androgen blockers or estradiol; no current or past exposure to androgen blockers or estradiol AND had sex with a person with a penis in the last year

Exclusion Criteria:

* Younger than 18 years old or older than 70 years old.
* Self-reported or documented history of nine-valent HPV vaccine or unsure of vaccination status and born after 2003.
* Born female
* History of hypersensitivity, including severe reactions to yeast or other component of the vaccine.
* Any condition requiring systemic chemotherapy or immunomodulant affecting antibody responses (i.e., rituximab, ibrutinib etc.), intravenous or subcutaneous immunoglobulin supplementation, radiation therapy, or immunomodulatory treatment within the previous 6 months (presence of precancerous lesions is not exclusionary).

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of the human papillomavirus (HPV) vaccine in BM-EABE (people born male with current or past exposure to androgen blockers or estrogen (BM-EABE) with and without HIV | 7 months post 1st vaccine dose
  Proportion of BM-EABE who become seropositive or have an increase in their GMT by >25% to at least 1 homologous HPV vaccine genotype at 1 month following the 3rd dose of the vaccine.

SECONDARY OUTCOMES:
Compare the humoral immune response to Gardasil9 between HIV positive BM-EABE and HIV negative controls | 7 months post 1st vaccine dose
  The difference between GMT titers against the 9-specific HPV types included in Gardasil between HIV positive BM-EABE and HIV negative controls.
Compare the humoral immune response to Gardasil9 between BM-EABE (regardless of HIV status) and BM without EABE (people born male without current or past exposure to androgen blockers or estrogen) | 7 months post 1st vaccine dose
  The difference between GMT titers against the 9-specific HPV types included in Gardasil between BM-EABE and BM without EABE
Evaluate the systemic HPV T-cell immune response to Gardasil9 in HIV positive BM-EABE and HIV negative controls. | 7 months post 1st vaccine dose
  A comprehensive assessment of HPV-specific T cell responses will be conducted with antigen stimulation of peripheral blood mononuclear cells (PBMCs) with virion-like protein (VLP) included in Gardasil 9. The proportion of proliferating T- cells, expressing activation-induced markers (AIM+) and IFN-gamma and TNF-alpha secreting T-cells will be evaluated by flow-cytometric assays; in addition the expression of exhaustion markers, perforin/granzyme B and skin- and gut-homing receptors, as well as the transcriptional analysis of T cells proliferating upon HPV antigenic stimulation will be assessed. This response will be assessed in HIV positive BM-EABE and HIV negative controls (BM-EABE and BM without EABE).
Compare systemic HPV T-cell immune response to Gardasil9 between HIV positive BM-EABE and HIV negative controls. | 7 months post 1st vaccine dose
  The proportion of proliferating T- cells, expressing activation-induced markers (AIM+) and IFN-gamma and TNF-alpha secreting T-cells, the expression of exhaustion markers, perforin/granzyme B and skin- and gut-homing receptors and the transcriptional analysis of T cells proliferating upon HPV antigenic stimulation will be compared between: HIV positive BM-EABE and HIV negative controls; BM-EABE and BM without EABE
Compare systemic HPV T-cell immune response to Gardasil9 between BM-EABE (regardless of HIV status) and BM without EABE. | 7 months post 1st vaccine dose
  The proportion of proliferating T- cells, expressing activation-induced markers (AIM+) and IFN-gamma and TNF-alpha secreting T-cells, the expression of exhaustion markers, perforin/granzyme B and skin- and gut-homing receptors and the transcriptional analysis of T cells proliferating upon HPV antigenic stimulation will be compared in BM-EABE and BM without EABE.
Evaluate the impact of HPV vaccination on HIV reservoir in CD4 T cells of BM-EABE with HIV. | Before vaccination, 7 months post 1st dose
  Distribution and density of mucosal immune cells (CD4+ and CD8+ T-cells, B/plasma cells, Dendritic/Langerhans cells, Natural killer (NK) cells, and macrophages) as seen on confocal microscopy from anal biopsies from HIV positive BM-EABE and HIV negative controls before Gardasil vaccination. Difference in distribution of mucosal immune cells as seen on confocal microscopy from anal biopsies after Gardasil.
Compare humoral immune response to Gardasil9 between different subset populations from PROTECT (HIV positive BM-EABE , HIV negative BM-EABE , and HIV negative MSPP), to age-matched historical controls. | 7 months post 1st vaccine dose
  The difference between GMT titers against the 9-specific HPV types included in Gardasil between subset of populations from PROTECT (HIV positive BM-EABE, HIV negative BM-EABE, men who have sex with a person with a penis (MSPP)) and historical controls from stored samples at the NIH

CONTACTS AND LOCATIONS:
Overall Officials: Omar Harfouch, MD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - RIIS Clinic at HIPS, Washington D.C., District of Columbia
  - RIIS Clinic at Baltimore Safe Haven, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator will share de-identified data with approved researchers at the time of publication or shortly afterwards.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of publication or shortly following publication, and will be available indefinitely.
Access Criteria: The criteria will be determined by the Principal Investigator